CLINICAL TRIAL: NCT01767103
Title: An Open-Label Study to Compare the Pharmacokinetic Profiles of a Single Dose of Ferriprox® in Subjects With Impaired Hepatic Function and Healthy Volunteers
Brief Title: An Open-label, Non-randomized, Parallel Group Study in Subjects With Mild and Moderate Hepatic Insufficiency and Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: LA40-0412
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Liver Impairment; Liver Disease; Ferriprox®; LI; DFP; Deferiprone
MeSH Terms: conditions — Liver Diseases | interventions — Deferiprone; Isoflurophate; Long Interspersed Nucleotide Elements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Hepatic Function (healthy volunteers) (Experimental): Healthy volunteers with normal hepatic function received a single 33 mg/kg dose of Ferriprox®.
  Interventions: Drug: Ferriprox®
- Mild Hepatic Failure (Experimental): Subjects with mild hepatic failure as defined by the Child-Pugh Class C: 5-6 points received a single 33 mg/kg dose of Ferriprox®.
  Interventions: Drug: Ferriprox®
- Moderate Hepatic Failure (Experimental): Subjects with moderate hepatic failure as defined by the Child-Pugh Class B: 7-9 points received a single 33 mg/kg dose of Ferriprox®.
  Interventions: Drug: Ferriprox®

INTERVENTIONS:
Drug: Ferriprox®
  Other Names: DFP; Deferiprone; L1

SUMMARY:
Multi-center, non-randomized, open-label, single-dose, parallel group study to determine the effect of impaired hepatic function on the PK of deferiprone and its 3-O-glucuronide metabolite following a single oral dose of 33mg/kg Ferriprox®.

DETAILED DESCRIPTION:
Post-marketing study to evaluate the effect of impaired hepatic function on the pharmacokinetics (PK) of deferiprone and its 3-O-glucuronide metabolite and on the safety of Ferriprox® in subjects with mild and moderate hepatic impairment as compared to healthy volunteers.

ELIGIBILITY:
Main Inclusion Criteria:

All subjects:

1. Adult males or females, 18 - 75 years of age (inclusive);
2. Body weight ≥ 50 kg;
3. Body mass index (BMI) between 19 and 32 kg/mE2 (inclusive);
4. Absolute neutrophil count (ANC) of >1.5x10E9/L ;

Healthy volunteers:

1. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical history, vital signs, physical examination);
2. Matched to hepatically impaired subjects in the study by age (+/- 10 years), sex and weight (+/- 15% BMI).

Hepatically impaired subjects:

1. Considered clinically stable in the opinion of the Investigator;
2. Subjects with different degrees of impaired hepatic function as assessed by a Child-Pugh classification score: mild (Class A: 5-6 points) and moderate (Class B: 7-9 points) impaired hepatic function.

Main Exclusion Criteria:

1. For subjects with hepatic impairment, fluctuating or rapidly deteriorating hepatic function as indicated by clinical and/or laboratory signs of hepatic impairment (e.g. advanced ascites, infection of ascites, fever, or active gastrointestinal bleeding).
2. Evidence of liver impairment in healthy volunteers: hepatitis B and C; or aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, clotting factors, serum protein that is considered clinically significant by the Investigator;
3. History or presence of significant clinically unstable respiratory, cardiovascular, pulmonary, hepatic (except for subjects assigned to one of the hepatically impaired groups), renal, hematologic, gastrointestinal, endocrine (except for subjects with hepatic impairment with clinically stable and treated diabetes, hypertension and thyroid disorders), immunologic, dermatologic, neurologic, or psychiatric disease;
4. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the PK of the investigational medicinal product (e.g. resections of the small or large intestine, febrile conditions, chronic diarrhea, chronic vomiting, clinically unstable endocrine disease, severe infections, acute inflammations, etc.);
5. Received a pharmacological agent in another clinical trial within 28 days prior to the first dose of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function (Healthy Volunteers): Healthy volunteers with normal hepatic function. All subjects received a single 33 mg/kg oral dose of deferiprone.
- Mild Hepatic Failure: Mild hepatic impairment as defined by Child-Pugh Class C: 5-6 points. All subjects received a single 33 mg/kg oral dose of deferiprone.
- Moderate Hepatic Failure: Moderate hepatic impairment as defined by Child-Pugh Class : 7-9 points. All subjects received a single 33 mg/kg oral dose of deferiprone.
Period: Overall Study
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Hepatic Function (Healthy Volunteers): Healthy volunteers with normal hepatic function
- Mild Hepatic Failure: Mild hepatic failure as defined by Child-Pugh Class C: 5-6 points
- Moderate Hepatic Failure: Moderate hepatic failure as defined by Child-Pugh Class B: 7-9 points
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 7 | 20
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 5
  Male | 5 | 7 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 6 | 7 | 6 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Cmax was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in subjects with normal hepatic function, mild hepatic impairment, or moderate hepatic impairment. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24-hour interval
Population: The PK Analysis Set consisted of all subjects who had sufficient data to derive at least one PK parameter
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Moderate Hepatic Failure: Moderate hepatic failure as defined by the Child-Pugh Class B: 7-9 points
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 7
ug/mL
  Cmax for serum deferiprone | 49.00 (24.081) | 36.26 (8.4799) | 35.94 (7.8407)
  Cmax for serum deferiprone 3-O-glucuronide | 69.03 (9.9153) | 56.91 (11.416) | 55.33 (25.335)

2. Secondary Outcome: Safety and Tolerability of Ferriprox in Subjects With or Without Hepatic Impairment.
Description: The number of participants who experienced adverse events following a single dose of Ferriprox, between the time of dosing and the follow-up visit (including any changes of clinical significance in physical examinations, vital signs, 12-lead ECG, and clinical laboratory tests).
Time Frame: Time of dosing until 48 hours post-dose
Population: The Safety Analysis Set consisted of all subjects who received study medication and had at least one safety assessment
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 7
participants | 0 | 1 | 3

3. Primary Outcome: Tmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Tmax was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in subjects with normal hepatic function, mild hepatic impairment, or moderate hepatic impairment. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24-hour interval
Population: The PK Analysis Set consisted of all subjects who had sufficient data to derive at least one PK parameter
Measure: Median (Full Range); unit: hour
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 7
hour
  Tmax of deferiprone | 0.7500 [0.500 to 2.00] | 0.7500 [0.500 to 1.00] | 0.7500 [0.500 to 1.33]
  Tmax of deferiprone 3-O-glucuronide | 2.000 [1.00 to 3.00] | 3.000 [1.67 to 4.00] | 3.000 [3.00 to 4.00]

4. Primary Outcome: AUC0-∞ for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUC (area under the curve) from zero to infinity was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in subjects with normal hepatic function, mild hepatic impairment, or moderate hepatic impairment. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24-hour interval
Population: The PK Analysis Set consisted of all subjects who had sufficient data to derive at least one PK parameter
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 7
ug*hr/mL
  AUC0-∞ for serum deferiprone | 92.64 (19.221) | 82.02 (28.213) | 105.5 (41.684)
  AUC0-∞ for serum deferiprone 3-O-glucuronide | 337.3 (45.343) | 305.1 (53.651) | 305.9 (111.75)

5. Primary Outcome: T1/2 for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: T1/2 was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in subjects with normal hepatic function, mild hepatic impairment, or moderate hepatic impairment. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24-hour interval
Population: The PK Analysis Set consisted of all subjects who had sufficient data to derive at least one PK parameter
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 7
hour
  T1/2 for serum deferiprone | 1.994 (0.26971) | 1.855 (0.45370) | 2.180 (0.83153)
  T1/2 for deferiprone 3-O-glu | 2.621 (0.35653) | 2.518 (0.55679) | 2.479 (0.67212)

6. Primary Outcome: CumAe for Urine Deferiprone and Deferiprone 3-O-glucuronide
Description: Cumulative amount of deferiprone and deferiprone 3-O-glucuronide excreted in the urine. Urine samples were collected at the intervals of -2 to 0 hours pre-dose, and 0-2, 2-4, 4-8, 8-12 ,and 12- 24 hours post-dose.
  Note: For unknown reasons, the urine samples for one subject in the moderate hepatic failure group had low or zero volume and there were no measurable levels of deferiprone or its metabolite in any of the samples. Accordingly, the urine PK results were derived both with and without this subject's data, and are here presented without them (i.e., N=6 rather than 7).
Time Frame: 24-hour interval
Population: The PK Analysis Set consisted of all subjects who had sufficient data to derive at least one PK parameter. The data of one subject in the moderate hepatic failure group were dropped due to low or zero volume of urine samples.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 6
mg
  CumAe of urine deferiprone | 69.0 (25.9) | 59.5 (19.4) | 62.9 (31.1)
  CumAe of urine deferiprone 3-O-glucuronide | 6670 (2520) | 6787 (619) | 5979 (887)

7. Primary Outcome: Fe% for Urine Deferiprone and Deferiprone 3-O-glucuronide
Description: Cumulative fraction of Ferriprox dose excreted in urine as deferiprone or deferiprone 3-O-glucuronide. Urine samples were collected at the intervals of -2 to 0 hours pre-dose, and 0-2, 2-4, 4-8, 8-12 ,and 12- 24 hours post-dose.
  Note: For unknown reasons, the urine samples for one subject in the moderate hepatic failure group had low or zero volume and there were no measurable levels of deferiprone or its metabolite in any of the samples. Accordingly, the urine PK results were derived both with and without this subject's data, and are here presented without them (i.e., N=6 rather than 7).
Time Frame: 24-hour interval
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of dose excreted in urine
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Number analyzed (Participants) | 7 | 7 | 6
percentage of dose excreted in urine
  Fe of urine deferiprone | 2.56 (0.773) | 2.18 (0.669) | 2.36 (1.20)
  Fe of urine 3-O-glucuronide | 109 (32.4) | 110 (14.0) | 97.7 (13.7)

ADVERSE EVENTS:
Time Frame: 2 days
Description: Safety data were collected from the time of dosing up to the follow-up visit 48 hours post-dose
Groups:
- Mild Hepatic Failure: Mild hepatic failure as defined by the Child-Pugh Class C: 5-6 points
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Hepatic Failure | Moderate Hepatic Failure
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (Healthy Volunteers) (N=7) | Mild Hepatic Failure (N=7) | Moderate Hepatic Failure (N=7)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (Healthy Volunteers) (N=7) | Mild Hepatic Failure (N=7) | Moderate Hepatic Failure (N=7)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retained title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the trial. Such publications shall not be made without the prior written consent of Sponsor. Neither Party will use the other Party's name in connection with any publication or promotion without the other Party's prior written consent. However, Sponsor has the right to publish appropriate information in order to satisfy regulatory requirements.